CLINICAL TRIAL: NCT05923073
Title: A Phase 3, Multicenter, Randomized, Platform Study of p19 Inhibition of the IL-23 Pathway to Establish Efficacy in Pediatric Crohn's Disease
Brief Title: A Study of Guselkumab in Pediatric Participants With Moderately to Severely Active Crohn's Disease
Acronym: MACARONI-23
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109212; CNTO1959PBCRD3007 (Other: Janssen Research & Development, LLC); 2021-006282-37 (EudraCT Number); 2023-504735-41-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
Keywords: Pediatric, Inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Open-label induction phase: Guselkumab Intravenously (IV) (Experimental): Participants will receive guselkumab dose IV based on their body weight during the 12-week open-label induction phase.
  Interventions: Drug: Guselkumab
- Open-label induction phase: Guselkumab Subcutaneously (SC) (Experimental): Participants will receive guselkumab dose SC based on their body weight during the 12-week open-label induction phase.
  Interventions: Drug: Guselkumab
- Double-blind maintenance phase: Guselkumab SC Dose Regimen 1 (Experimental): At the end of the induction phase, Week 12 responders will be randomized into the double-blind maintenance phase to receive guselkumab dose regimen 1 SC based on their body weight up to Week 48.
  Interventions: Drug: Guselkumab
- Double-blind Maintenance Phase: Guselkumab SC Dose Regimen 2 (Experimental): At the end of the induction phase, Week 12 responders will be randomized into the double-blind maintenance phase to receive guselkumab dose regimen 2 SC based on their body weight up to Week 48.
  Interventions: Drug: Guselkumab
- Open-label maintenance phase: Guselkumab SC (Experimental): Week 12 non-responders will not be randomized and will enter an open-label maintenance phase to receive guselkumab SC dosing regimen based on their body weight up to Week 48.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously.
  Other Names: CNTO1959; TREMFYA
  Arms: Double-blind Maintenance Phase: Guselkumab SC Dose Regimen 2; Double-blind maintenance phase: Guselkumab SC Dose Regimen 1; Open-label induction phase: Guselkumab Subcutaneously (SC); Open-label maintenance phase: Guselkumab SC
Drug: Guselkumab — Guselkumab will be administered intravenously.
  Other Names: CNTO1959; TREMFYA
  Arms: Open-label induction phase: Guselkumab Intravenously (IV)

SUMMARY:
The purpose of this study is to evaluate the clinical and endoscopic efficacy of guselkumab in pediatric participants with Crohn's Disease (CD) at the end of maintenance therapy (Week 52) among participants who were in clinical response to guselkumab at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of Crohn's Disease (CD) or fistulizing CD, with active colitis, ileitis, or ileocolitis, confirmed at any time in the past by clinical, endoscopic, and histologic criteria.
* Participants must have moderately to severely active CD (as defined by a baseline Pediatric Crohn's Disease Activity Index [PCDAI] score greater than or equal to [>=] 30)
* Participants must have endoscopy with evidence of active CD defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) score greater than or equal to (>=) 6 (or >=4 for participants with isolated ileal disease) within 1 month of receiving study intervention at Week 0
* Participants must have a history of inadequate response, loss of response, or intolerance to immunomodulators (6-MP, AZA, or MTX), oral or IV corticosteroids, or biologic therapy/JAK inhibitor therapy; OR have a history of corticosteroid dependence; OR have a history of inadequate response to exclusive enteral nutrition (EEN)

Exclusion Criteria:

* Participants has complications of CD such as symptomatic strictures or stenosis, short gut syndrome, or any other manifestation that might be anticipated to require surgery.
* Participants must not have an abscess
* Participants must not have any kind of bowel resection within 26 weeks or any other intra-abdominal surgery within 12 weeks of baseline

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-10-27 (Estimated); Study Completion 2028-07-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 52 | Week 52
  Percentage of participants with clinical remission at Week 52 will be assessed. Clinical remission is defined as pediatric Crohn's Disease activity index (PCDAI) less than or equal to (<=) 10.
Percentage of Participants Who Achieve Endoscopic Response at Week 52 | Week 52
  Percentage of participants who achieve endoscopic response at Week 52 will be assessed. Endoscopic response is defined as greater than or equal to (>=) 50 percent (%) reduction (global) and greater than (>) 50% reduction (U.S specific) from simplified endoscopic score-Crohn's Disease (SES-CD) score at baseline.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 12 | Week 12
  Percentage of participants with clinical response at Week 12 will be assessed. Clinical responder is defined as a decrease from baseline in the PCDAI score of >=12.5 points with a total PCDAI score <30.
Percentage of Participants with Clinical Response at Week 52 | Week 52
  Percentage of participants with clinical response at Week 52 will be assessed. Clinical responder is defined as a decrease from baseline in the PCDAI score of >=12.5 points with a total PCDAI score <30.
Percentage of Participants with Clinical Remission at Week 12 | Week 12
  Percentage of participants with clinical remission at Week 12 will be assessed. Clinical remission is defined as PCDAI score <=10.
Percentage of Participants with Endoscopic Remission at Week 52 | Week 52
  Percentage of participants with endoscopic remission at Week 52 will be assessed. Endoscopic remission is defined as SES-CD total score <=4 and at least a 2-point reduction from baseline and no subscore >1.
Percentage of Participants with Corticosteroid-free Remission at Week 52 | Week 52
  Percentage of participants with corticosteroid-free remission at Week 52 will be assessed. Corticosteroid-free remission is defined as PCDAI score <=10 at Week 52 and not receiving corticosteroids for at least 90 days before Week 52.
Percentage of Participants with Sustained Clinical Remission at Weeks 12, 24, and 52 | Weeks 12, 24, and 52
  Percentage of participants with sustained clinical remission at Weeks 12, 24, and 52 will be assessed. Sustained clinical remission is defined as PCDAI <=10 at Weeks 12, 24, and 52.
Percentage of Participants with Clinical remission by Patient-Reported Outcome (PRO-2) | Week 12 and/or Week 52
  Percentage of participants with clinical remission by PRO-2 will be assessed. Clinical remission by PRO-2 is defined as stool frequency (SF) <=3 and abdominal pain (AP) <=1 and no worsening of SF and AP from baseline.
Serum Concentration of Guselkumab During Induction Phase | From Week 0 to Week 12
  Serum concentrations of guselkumab will be assessed. Serum samples will be analyzed to determine concentrations of guselkumab using a validated, specific, and sensitive immunoassay method.
Trough Plasma Concentration (Ctrough) of Guselkumab During Maintenance Phase | At Weeks 16, 24, 36, 48 and 52
  Ctrough is defined as the serum concentration of guselkumab immediately prior (pre-dose) to the next drug administration.
Change from Baseline in Body Weight at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in body weight at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Body Weight Percentiles at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in body weight percentiles at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Body Weight z-scores at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in body weight z-scores at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Height at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in height at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Height Percentiles at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in height percentiles at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Height z-scores at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in height z-scores at Weeks 12, 24, and 52 will be assessed.
Change from Baseline in Height Velocity at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
  Change from baseline in height velocity at Weeks 12, 24, and 52 will be assessed.
Percentage of Participants with Clinical Remission | Week 52
  Percentage of participants with clinical remission who were assigned to guselkumab dose regimen 1 and did not receive rescue therapy at Week 52 will be assessed. Clinical remission is defined as PCDAI score <=10.
Percentage of Participants Who Achieve Endoscopic Response | Week 52
  Percentage of participants who achieve endoscopic response who were assigned to q4w maintenance therapy and did not receive rescue therapy at Week 52 will be assessed. Endoscopic response is defined as >=50% reduction (global) and >50% reduction (U.S specific) from SES-CD score at baseline.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 64
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. An SAE is is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (79):
- United States (13):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Childrens Hospital, Boston, Massachusetts
  - Weill Cornell Medical College - Judith Jaffe Multiple Sclerosis Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Childrens Medical Center, Fort Worth, Texas
  - University of Vermont Medical Center, Colchester, Vermont
- Australia (2):
  - Mater Hospital Brisbane, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- AKH - Medizinische Universitat Wien, Vienna, Austria
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (7):
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Associacao Hospitalar de Protecao a Infancia Dr. Raul Carneiro, Curitiba
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Centro de Ciencias e Saude da Universidade Federal do Espirito Santo-Nucleo de Doencas Infecciosas, Vitória
  - INTEGRAL Pesquisa e Ensino, Votuporanga
- Canada (2):
  - Iwk Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre Victoria Hospital, London, Ontario
- France (4):
  - CHU Amiens-Hopital Nord, Amiens
  - Hôpital Jeanne de FLANDRE, CHRU LILLE, Lille
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Ospedale Bellaria, U.O.Cardiologia Az. USL di Bologna, Bologna
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Presidio Ospedale dei Bambini Vittore Buzzi, Milan
  - AOU Policlinico Umberto I, Roma
- Japan (10):
  - Hirosaki University Hospital, Hirosaki
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi
  - Kobe University Hospital, Kobe
  - Saga University Hospital, Saga
  - Miyagi Children's Hospital, Sendai
  - National Center for Child Health and Development, Setagaya Ku
  - Juntendo University Hospital, Tokyo
  - Mie University Hospital, Tsu
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Norway (4):
  - Akershus Universitetssykehus HF, Nordbyhagen
  - Oslo University Hospital, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - St. Olavs Hospital, Trondheim
- Poland (3):
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut Pomnik Centrum Zdrowia, Warsaw
- Portugal (3):
  - Hospital de Braga, Braga
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - Centro Hospitalar de Sao Joao E.P.E., Porto
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (3):
  - Hosp Reina Sofia, Córdoba
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. I Politecni La Fe, Valencia
- United Kingdom (6):
  - Royal Hospital for Sick Children, Glasgow
  - Great Ormond Street Hospital, London
  - Nowgen Centre, Research and Innovation, Manchester
  - Royal Manchester Children's Hospital, Manchester
  - John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency